CLINICAL TRIAL: NCT02422563
Title: Multicenter Prospective Randomized Study on NeoAdjuvant Chemotherapy Followed by Radical Hysterectomy (OP) Versus Primary Chemo-RADiation in Patients With Cervical Cancer FIGO Stage IB2 and IIB
Brief Title: NeoAdjuvant Chemotherapy Followed by Radical Hysterectomy (OP) Versus Primary Chemo-RADiation in Cervical Cancer FIGO Stage IB2 and IIB
Acronym: NACOPRAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, S. Marnitz, Prof. Dr. med. S. Marnitz, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NACOPRAD_2015
Record Dates: First submitted 2015-02-11; First posted 2015-04-21 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Cervical Cancer
Keywords: neoadjuvant chemotherapy; FIGO IB2, FIGO IIB; chemo-radiation; dose dense chemotherapy; cisplatin; paclitaxel; carboplatin; ifosfamide
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Hysterectomy; Radiation; Cisplatin; Paclitaxel; Carboplatin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: NACT+radical hysterectomy (Experimental): Arm A includes patients for dose dense chemotherapy using TP (paclitaxel, carboplatin) or TIP (cisplatin, paclitaxel, ifosfamide) weekly for six cycles. Radical hysterectomy is performed after the 6th week + lymphadenectomy
  Interventions: Procedure: hysterectomy; Drug: Cisplatin; Drug: Paclitaxel; Drug: Carboplatin; Drug: Ifosfamide
- Arm B: Chemoradiation (Other): Arm B includes patients undergoing primary cisplatin based chemo-radiation
  Interventions: Radiation: Radiation; Drug: Cisplatin

INTERVENTIONS:
Procedure: hysterectomy — radical hysterectomy
  Arms: Arm A: NACT+radical hysterectomy
Radiation: Radiation
  Arms: Arm B: Chemoradiation
Drug: Cisplatin
Drug: Paclitaxel
  Arms: Arm A: NACT+radical hysterectomy
Drug: Carboplatin
  Arms: Arm A: NACT+radical hysterectomy
Drug: Ifosfamide
  Arms: Arm A: NACT+radical hysterectomy

SUMMARY:
Randomized comparison of neoadjuvant chemotherapy followed by radical hysterectomy with pelvic ± para-aortic lymphonodectomy (LNE) versus primary cisplatin-based chemo-radiation in patients with cervical cancer FIGO IB2 and IIB.

DETAILED DESCRIPTION:
The optimal treatment for patients with cervical cancer on FIGO stage IB2 and IIB is controversial. There is no randomized comparison of a dose-dense NACT (TP or TIP-schedule) followed by hysterectomy and LNE (investigational Arm A) versus primary chemo-radiation (standard arm B). Primary endpoint is the DFS at 5 years, secondary endpoints local control at 5 years, OS at 5 years, QOL, questionnaires on sexual activity/QOL.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* cervical cancer FIGO IB2, IIB,
* squamous cell, adeno or adenosquamous cell carcinoma
* informed consent

Exclusion Criteria:

* small cell/neuroendocrine component
* previous radiation, previous cancer
* pregnancy
* HIV
* severe co-morbidities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years
  DFS

SECONDARY OUTCOMES:
overall survival | 5 years
local control | 5 years
  local control rate at 5 years
quality of life | 5 years
  Qol questionnaire EORTC Qol C30 and Cervical Cancer Module EORTC QLQ-CX24

REFERENCES:
- [Background] Sardi JE, di Paola GR, Cachau A, Ortiz OC, Sananes C, Giaroli A, Martins D, Peluffo M. A possible new trend in the management of the carcinoma of the cervix uteri. Gynecol Oncol. 1986 Oct;25(2):139-49. doi: 10.1016/0090-8258(86)90095-8. PMID 2428700
- [Background] Benedetti-Panici P, Greggi S, Colombo A, Amoroso M, Smaniotto D, Giannarelli D, Amunni G, Raspagliesi F, Zola P, Mangioni C, Landoni F. Neoadjuvant chemotherapy and radical surgery versus exclusive radiotherapy in locally advanced squamous cell cervical cancer: results from the Italian multicenter randomized study. J Clin Oncol. 2002 Jan 1;20(1):179-88. doi: 10.1200/JCO.2002.20.1.179. PMID 11773168
- [Background] Sardi J, Sananes C, Giaroli A, Maya G, di Paola G. Neoadjuvant chemotherapy in locally advanced carcinoma of the cervix uteri. Gynecol Oncol. 1990 Sep;38(3):486-93. doi: 10.1016/0090-8258(90)90096-4. PMID 1699851
- [Background] Souhami L, Gil RA, Allan SE, Canary PC, Araujo CM, Pinto LH, Silveira TR. A randomized trial of chemotherapy followed by pelvic radiation therapy in stage IIIB carcinoma of the cervix. J Clin Oncol. 1991 Jun;9(6):970-7. doi: 10.1200/JCO.1991.9.6.970. PMID 1709686
- [Background] Gadducci A, Sartori E, Maggino T, Zola P, Cosio S, Zizioli V, Lapresa M, Piovano E, Landoni F. Pathological response on surgical samples is an independent prognostic variable for patients with Stage Ib2-IIb cervical cancer treated with neoadjuvant chemotherapy and radical hysterectomy: an Italian multicenter retrospective study (CTF Study). Gynecol Oncol. 2013 Dec;131(3):640-4. doi: 10.1016/j.ygyno.2013.09.029. Epub 2013 Oct 3. PMID 24096111
- [Background] Lissoni AA, Colombo N, Pellegrino A, Parma G, Zola P, Katsaros D, Chiari S, Buda A, Landoni F, Peiretti M, Dell'anna T, Fruscio R, Signorelli M, Grassi R, Floriani I, Fossati R, Torri V, Rulli E. A phase II, randomized trial of neo-adjuvant chemotherapy comparing a three-drug combination of paclitaxel, ifosfamide, and cisplatin (TIP) versus paclitaxel and cisplatin (TP) followed by radical surgery in patients with locally advanced squamous cell cervical carcinoma: the Snap-02 Italian Collaborative Study. Ann Oncol. 2009 Apr;20(4):660-5. doi: 10.1093/annonc/mdn690. Epub 2009 Jan 30. PMID 19181826
- [Background] Buda A, Fossati R, Colombo N, Fei F, Floriani I, Gueli Alletti D, Katsaros D, Landoni F, Lissoni A, Malzoni C, Sartori E, Scollo P, Torri V, Zola P, Mangioni C. Randomized trial of neoadjuvant chemotherapy comparing paclitaxel, ifosfamide, and cisplatin with ifosfamide and cisplatin followed by radical surgery in patients with locally advanced squamous cell cervical carcinoma: the SNAP01 (Studio Neo-Adjuvante Portio) Italian Collaborative Study. J Clin Oncol. 2005 Jun 20;23(18):4137-45. doi: 10.1200/JCO.2005.04.172. PMID 15961761
- [Background] Landoni F, Sartori E, Maggino T, Zola P, Zanagnolo V, Cosio S, Ferrari F, Piovano E, Gadducci A. Is there a role for postoperative treatment in patients with stage Ib2-IIb cervical cancer treated with neo-adjuvant chemotherapy and radical surgery? An Italian multicenter retrospective study. Gynecol Oncol. 2014 Mar;132(3):611-7. doi: 10.1016/j.ygyno.2013.12.010. Epub 2013 Dec 14. PMID 24342439